CLINICAL TRIAL: NCT05536258
Title: Evaluation of the ZYNEX Cardiac Monitor in Patients Having Noncardiac Surgery
Brief Title: ZYNEX Cardiac Monitor in Patients Having Noncardiac Surgery
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 22-340
Record Dates: First submitted 2022-09-07; First posted 2022-09-10 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Noncardiac Surgery
MeSH Terms: interventions — Fluid Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- RI-Monitoring: The investigator will evaluate the feasibility of a RI-guided fluid ministration for improving perioperative characteristics.
  Feasibility will be defined by:
  The investigators will titrate fluid administration to maintain a RI > 90 over at least 85% of the intraoperative period lasting from induction until the end of anesthesia. Specifically, the investigator will consider titration to have been successful if 85% of patients in the RI group sustain a RI > 90 over at least 85% of the intraoperative period;
  Interventions: Other: Fluid

INTERVENTIONS:
Other: Fluid — The investigators will titrate fluid administration to maintain a RI > 90 over at least 85% of the intraoperative period lasting from induction until the end of anesthesia. Specifically, the investigator will consider titration to have been successful if 85% of patients in the RI group sustain a RI > 90 over at least 85% of the intraoperative period.

SUMMARY:
The trial groups will be:

1. Routine fluid management. Clinicians will be blinded to RI monitoring and use clinical judgement to determine how much fluids should be given, and when. Clinical judgement will be according to their standard practice and may include interpretation of blood pressure, and heart rate.
2. RI-guided fluid administration. RI fluid guidance will be initiated before anesthesia induction and will maintain until end of anesthesia. Clinicians will titrate fluids with the goal of keeping RI above 90- always using good clinical judgement for individual patients which may include avoiding fluid when RI is <90 or giving additional fluid when RI >90. For RI scores below 90, 1 cc/kg actual body weight fluid bolus of any crystalloid solution (normal saline or Ringer's lactate) will be given; colloids and blood products can also be given if clinically indicated. The target will be maintained until end of anesthesia.

Anesthesia will be maintained for the entire surgical procedure per clinical routine. At the end of the surgical procedure, patients will be extubated and transferred to the post anesthesia care unit (PACU).

DETAILED DESCRIPTION:
Patients will be premedicated with 0-2 mg midazolam per preference of the attending anesthesiologist. General anesthesia will be induced as preferred by the attending anesthesiologist, usually with a combination of lidocaine 1 mg/kg, propofol 1-4 mg/kg, fentanyl 1-2 µg/kg, and rocuronium 0.6-1.2 mg/kg or succinylcholine 1.5 mg/kg. The trachea will be intubated, and the lungs mechanically ventilated per clinical routine. General anesthesia will be maintained with an initial sevoflurane target concentration of 0.8% which will be adjusted based on apparent clinical need, supplemented with fentanyl. Vasopressors, antihypertensives, and drugs to control heart rate may be given as clinically indicated. BIS will be recorded to estimate hypnotic depth.

Patients will be randomized 1:1, stratified for chronic use of antihypertensive medication, in random-sized blocks to RI-guided fluid management or routine care. The randomization table will be prepared by trial statisticians, and allocation will be concealed until shortly before anesthetic induction with a web-based randomization system. The Zynex RI system will be applied and calibrated before anesthetic induction in all patients. A continuous fluid infusion of 1cc/ kg actual body weight/hour of crystalloid solution will be started in all patients before anesthesia induction and maintained until end of anesthesia. The trial groups will be:

1. Routine fluid management. Clinicians will be blinded to RI monitoring and use clinical judgement to determine how much fluids should be given, and when. Clinical judgement will be according to their standard practice and may include interpretation of blood pressure, and heart rate.
2. RI-guided fluid administration. RI fluid guidance will be initiated before anesthesia induction and will maintain until end of anesthesia. Clinicians will titrate fluids with the goal of keeping RI above 90- always using good clinical judgement for individual patients which may include avoiding fluid when RI is <90 or giving additional fluid when RI >90. For RI scores below 90, 1 cc/kg actual body weight fluid bolus of any crystalloid solution (normal saline or Ringer's lactate) will be given; colloids and blood products can also be given if clinically indicated. The target will be maintained until end of anesthesia.

Anesthesia will be maintained for the entire surgical procedure per clinical routine. At the end of the surgical procedure, patients will be extubated and transferred to the post anesthesia care unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

1. Adults having major non-cardiac surgery expected to last ≥2 hours
2. American Society of Anesthesiologists physical status 1-3
3. Age 21-85 years old
4. Planned endotracheal intubation and general anesthesia with or without any regional blocks.

Exclusion Criteria:

1. Non-sinus heart rhythm;
2. amputation of any extremity;
3. eGFR < 30 including end-stage kidney disease;
4. cardiac ejection fraction < 50;
5. temporary or permanent pacemaker;
6. BMI > 40 kg/m2. -

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients having major non-cardiac surgery expected to last ≥2 hours. The ASA physical status 1-3, and their age 21-85 years old. The patient should have a planned endotracheal intubation and general anesthesia with or without any regional blocks.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Identify absolute and relative changes of RI | PACU stay
  continuously monitor and obtain RI values throughout anesthesia and the post anesthesia care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Ruetzler, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States